CLINICAL TRIAL: NCT05647863
Title: Improving Rehabilitation Compliance and Treatment Duration by Treating Executive Function and Sensory Modulation Deficits in Individuals With Substance Use Disorder: A Randomized Control Trial
Brief Title: F-CaST for Individuals With Substance Use Disorder
Acronym: F-CaST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel Aviv University (Other)
Responsible Party: Principal Investigator, Tami Bar-Shalita, Principal Investigator, Tel Aviv University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 0001484-4
Record Dates: First submitted 2022-08-10; First posted 2022-12-13 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Substance Use Disorders
Keywords: Rehabilitation compliance; Executive functions; Sensory modulation dysfunction
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with an experimental group and a control group
Who Masked: Outcomes Assessor
Masking Description: Assessors in the RCT will be blind to group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- F-CaST (Experimental): The experimental group who will receive the Functional Cognitive and Sensory Treatment (F-CaST)- in which therapy is individually tailored for successful task performance and where the focus is on strategies for improving sensory and EF deficits.
  Interventions: Other: Functional Cognitive and Sensory Treatment (F-CaST)
- Standard Care (No Intervention): Standard care at the therapeutic community for SUD.

INTERVENTIONS:
Other: Functional Cognitive and Sensory Treatment (F-CaST) — F-CaST, a client-centered care, is a functional cognitive sensory intervention focusing on improving Executive Function (EF) and sensory modulation impairments using a modification of the Functional and Cognitive Occupational Therapy Treatment.
  Other Names: Cognitive sensory occupational therapy
  Arms: F-CaST

SUMMARY:
Examining the effectiveness of the F-CaST based on a controlled randomized trial in patients with SUD residing in a therapeutic community.

DETAILED DESCRIPTION:
Background and Aims: Substance use disorder (SUD), an urgent public health concern, is a chronic relapsing brain disorder caused by psychoactive substances, characterized by cognitive, behavioral, and physiological symptoms, severely impacting every life domain. Repeated substance use leads to impairments in higher cognitive abilities, termed executive functions (EF), and leads to SUD chronicity. Furthermore, EF deficits are associated with difficulties in sensory processing, severely limiting daily functions and with reported high incidence in SUD. However, to date both are not addressed therapeutically. This translational study aims to enhance rehabilitation success in patients with SUD residing in a therapeutic community (TC) by employing sensory and EF strategies utilizing the Functional Cognitive and Sensory Treatment (F-CaST), an innovative personalized therapy.

Methods: A qualitative study will be nested in a single-blind, controlled randomized trial, comparing two groups: (i) Experimental group- F-CaST - in which therapy is individually tailored for successful task performance and where the focus is on strategies for improving sensory and EF deficits and (ii) Control group - Standard Care - the typical treatment given in the therapeutic community. Measurement will be conducted by assessors blind to group allocation at 4 time points: T1- pre-intervention; T2- post-intervention; T3- at a 1-month follow-up; and T4- at a 3-month follow-up.

Population: Forty-eight adults diagnosed with SUD, aged 18-45 years, with no significant cognitive deficits, and residing in a TC for SUD.

Tools: Both objective and subjective measures to evaluate TC performance will be applied. Additionally, interviews will be conducted to provide a deeper understanding of the perceived performance and difficulties.

Expected Results: F-CaST will lead to improved rehabilitation success and treatment duration, better compliance with TC requirements, and greater satisfaction, compared to control group.

ELIGIBILITY:
Inclusion criteria:

* Diagnosed by a psychiatrist and meeting the DSM-V diagnostic criteria for severe SUD
* Admitted to the therapeutic community (TC) for full-length SUD rehabilitation and with no more than 3 previous rehabilitation trials in this TC
* Abstained from drugs and alcohol for at least 14 days (verifying minimum withdrawal effects); and no more than 21 days of TC residency (to ensure familiarization with the facility)
* Without a significant cognitive deficit [the Montreal Cognitive Assessment (MoCA)≥19/30 points) and adequate language skills

Exclusion Criteria:

* Relapsing substance use in the TC

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2022-11-25 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Change The Canadian Occupational Performance Measure (COPM) | Change in The Canadian Occupational Performance Measure between pre (T1-week 0) to T2 (post-intervention 8-9 weeks later), to T3 (follow-up- one month later) and T4 (follow-up- three months later). Higher scores indicate better outcomes
  The Canadian Occupational Performance Measure (COPM) is a client-centered outcome measure for individuals to identify and prioritize everyday issues that restrict their participation in everyday living.
  Participants will define three goals, and rate their current performance & satisfaction for each goal using a 10-point scale. Higher scores indicate better outcomes.
Length of stay in Therapeutic Community | At T4 ( three months later after follow-up) or earlier (when they leave the TC)
  Length of stay (days) residing in Therapeutic Community. Longer time spent in the TC is better.
Change in Performance in the Therapeutic Community | Change in Performance in the Therapeutic Community between pre (T1-week 0) - to post (T2- post-intervention 8-9 weeks later) to T3 (follow-up- one month later) and T4 (follow-up- three months later).
  Participant performance in the Therapeutic Community will be based on the community counselor's evaluation. Better performance is better
Change in number of times coming late for scheduled appointments | Change in number of times coming late for scheduled appointments between pre (T1-week 0) - to post (T2- post-intervention 8-9 weeks later) to T3 (follow-up- one month later) and T4 (follow-up- three months later).
  Number of times coming late for scheduled appointments. Less times of coming late is better.

SECONDARY OUTCOMES:
Four Item Tablet Test (4ITT) | Change between pre (T1-week 0) to T2 (post-intervention 8-9 weeks later), T3 (follow-up- one month later) and T4 (follow-up- three months later)]
  Performance test of executive functioning via a quick online shopping task using a tablet.
  Scores will include shopping time & mistakes - less time with less mistakes is better shopping performance.
Color Trails Test (CTT) | Change between pre (T1-week 0) to T2 (post-intervention 8-9 weeks later), T3 (follow-up- one month later) and T4 (follow-up- three months later)]
  A pen and paper neuropsychological test used to measure cognitive flexibility and processing speed. The CTT includes two parts: (1) CTT part 1 requires to connect a series of 25 numbered circles that are scattered on a sheet of paper and (2) CTT part 2 requires to connect numbered circles from 1 to 25 in sequence alternating between two colors-pink and yellow (1-pink, 2-yellow, 3-pink, 4-yellow…). The time (seconds) to complete each part will be recorded. Completion time (up to 240 seconds) translated to standardized score by normative data correcting for age and years of education. The CTT is widely used in a variety of populations and was found as a valid and reliable measure with a variety of populations.
  Less time (secs) indicates better executive function.
Behavior Rating Inventory of Executive Function-Adult Version (BRIEF-A) | Change between pre (T1-week 0) to T2 (post-intervention 8-9 weeks later), T3 (follow-up- one month later) and T4 (follow-up- three months later)]
  A 75-item questionnaire assessing EF in everyday environments. BRIEF-A is composed of nine clinical scales which form two indices: (i) the Behavioral Regulations Index (BRI), and (ii) the Metacognition Index (MI). The BRI and MI together produce an overall Global Executive Composite (GEC). Based on the past 30 days, items are graded on a 3-point scale: 'never' (1), 'sometimes' (2), or 'always' (3). The raw scores are converted to T-scores where a score of 65 or higher denotes a clinical deficit. Higher scores indicate worse outcomes.
Computerized cognitive assessment battery (CANTAB) | Change between pre (T1-week 0) to T2 (post-intervention 8-9 weeks later), T3 (follow-up- one month later) and T4 (follow-up- three months later)]
  Two computerized tasks from the Cambridge Automatic Neuropsychological Test Battery (CANTAB) subtests will be used to assess multitasking and working memory.
  The tasks will be administered using a touchscreen tablet:
  The Multitasking Test (MTT) Spatial Working Memory (SWM)
The Self-Regulation Skills Interview | Change between pre (T1-week 0) to T2 (post-intervention 8-9 weeks later), T3 (follow-up- one month later) and T4 (follow-up- three months later)]
  A semi-structured interview composed of six questions that assess a range of metacognitive skills essential for rehabilitation planning, monitoring an individual's progress, and evaluating the outcome of treatment interventions. The six questions are applied to a main area of difficulty experienced in everyday living as identified by the individual.
The Sensory Responsiveness Questionnaire-Intensity Scale | Change between pre (T1-week 0) to T2 (post-intervention 8-9 weeks later), T3 (follow-up- one month later) and T4 (follow-up- three months later)]
  A 58-item questionnaire aimed at clinically classifying sensory modulation dysfunction in adults. Items represent typical daily life situations involving auditory, visual, gustatory, olfactory, vestibular and somatosensory sensations, excluding pain. Items are phrased either in a hedonic or aversive valence and are graded on a 5-point Likert scale: 'not at all' (1) to 'very much' (5). Two cut-off scores are provided.
The Pain Sensitivity Questionnaire | Change between pre (T1-week 0) to T2 (post-intervention 8-9 weeks later), T3 (follow-up- one month later) and T4 (follow-up- three months later)]
  A 17 item questionnaire aimed to quantify everyday somatosensory pain sensitivity to imagined painful daily life situations. Participants rate the intensity of imagined pain on a 10-point scale: 'not painful at all' (0) to 'the worst pain imaginable' (10). The Pain Sensitivity Questionnaire provides a total score and two sub-scores.
The New General Self-Efficacy Scale | Change between pre (T1-week 0) to T2 (post-intervention 8-9 weeks later), T3 (follow-up- one month later) and T4 (follow-up- three months later)]
  An 8-item measure that assesses how much people believe they can achieve their goals despite their difficulties. Each of the eight statements (e.g. "Even when things are tough, I can perform quite well") are rated using a 5-point rating scale: 'strongly disagree' (1) to 'strongly agree' (5); higher scores indicate higher self-efficacy.
Satisfaction with Life Scale | Change between pre (T1-week 0) to T2 (post-intervention 8-9 weeks later), T3 (follow-up- one month later) and T4 (follow-up- three months later)]
  A self-report questionnaire measuring global life satisfaction. This scale examines the cognitive component of subjective well-being and consists of five statements that reflect the overall satisfaction of an individual's life. Responders are asked to rate the level of agreement with each statement on a scale ranging from 1 (total disagreement) to 7 (total agreement). Higher scores indicate better life satisfaction.
In-depth semi-structured interview | Pre (T1-week 0), T2 (post-intervention 8-9 weeks later), T3 (follow-up- one month later) and T4 (follow-up- three months later)
  A semi-structured interview, comprising of 5 open-end questions aiming to understand how adults with SUD perceive their performance at the TC and the link between their performance to their executive functioning and sensory modulation disorder. The interview will comprise questions such as What, in your opinion, can explain your performance?
  Each time point will be analyzed separately.
The World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0) - 12 item version | Change between pre (T1-week 0) to T2 (post-intervention 8-9 weeks later), T3 (follow-up- one month later) and T4 (follow-up- three months later)
  Assesses activity limitations and participation restrictions in daily activities. The WHODAS 2.0 comprises six major life domains yielding the sub-scales: Cognition; Household (life activity); Mobility; Self-care; Social; and Participation in Society. Items are graded on a 5-point Likert scale: "none" (0) to "extreme" (4), where higher scores denote higher disability.

OTHER OUTCOMES:
Montreal Cognitive Assessment | T1- pre-intervention
  A 10-minute cognitive screening tool assessment for detecting cognitive impairment. The MoCA items include short term memory recall, visuospatial ability, executive function, attention-concentration-working memory, language, and orientation to time and place.
  Scores range from 0-30, higher scores indicate better cognition
The Adult ADHD Self-Report Scale-Version 1.1 | Change between pre (T1-week 0) to T2 (post-intervention 8-9 weeks later), T3 (follow-up- one month later) and T4 (follow-up- three months later)]
  A 18-item checklist for screening adult Attention deficit hyperactivity disorder based on the Diagnostic and Statistical Manual of Mental Disorders -IV diagnostic criteria using a 5 point Likert scale 'Never' (0) to 'Very Often' (4).
The Satisfaction from the intervention questionnaire | Post intervention (T2, which is 8-9 weeks after T1)
  A 9-item questionnaire measuring the patient satisfaction with the intervention.
  Higher scores - more satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Naama Assayag, Dr., Principal Investigator — Tel Aviv University
Locations (1):
- Malkishua, Afula, Israel

IPD SHARING:
Plan to Share IPD: No
Data will be available upon personal request

REFERENCES:
- [Derived] Assayag N, Bar-Shalita T, Rand D. The Functional-Cognitive and Sensory Treatment (F-CaST) to improve rehabilitation outcomes of individuals with substance use disorder: a study protocol for a mixed-method randomized controlled trial. Addict Sci Clin Pract. 2024 Apr 9;19(1):28. doi: 10.1186/s13722-024-00449-7. PMID 38594737